CLINICAL TRIAL: NCT05079594
Title: Investigation of Infant Comfort Levels and Mothers' Anxiety Levels in Non-pharmacological Maternal Voice and White Noise Methods in Heel Blood Procedure
Brief Title: The Effects of Auditory Interventions on Comfort and Mothers' Anxiety in Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Uğur Gül, Research Assistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Akdeniz Faculty of Nursing
Record Dates: First submitted 2021-10-04; First posted 2021-10-15 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Pain, Acute
Keywords: white noise; pain; Mother's voice; pain management; newborn
MeSH Terms: conditions — Acute Pain; Pain; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Routine Care Group (No Intervention): Before the application, the families will be informed by the researcher and the 'Informed Consent Form' will be signed. After the heel blood procedure, when the baby starts to cry, comfort will be provided with gentle touches. For ethical reasons, routine care will be provided when the baby cries.
- White Noise (Experimental): Since white noise is a humming and continuous monotonous sound, it is similar to the sound in the womb. It will be explained that this sound is very similar to the sound that the baby hears in the mother's womb by making the white noise recordings listen to the mothers who will have their babies listen to white noise. by Orhan Osman; Dr. From the album 'Kolik', which was created by making use of the album 'The Happiest Baby' prepared by Harvey Karp, which consists only of uterus sounds; The song 'Don't Let Your Baby Cry, PT.2' will be played to babies. In addition, infants will be excluded from the study even though they meet the criteria, if they are not sedated, the procedure takes more than 2 minutes, the procedure is disrupted because someone enters the room loudly, or the mother changes the baby's position.
  Interventions: Other: White noise
- Mother Voice (Experimental): Auditory responses, fetal age 26-28. It develops in the auditory cortex and brain stem in weeks. Hearing is one of the first senses a fetus develops and is 24-33. can recognize and remember the mother's voice after weeks. The fetus memorizes the musical characteristics of the mother's voice, like tone, by listening to it. It is stated that newborns exposed to their own mother's voice have a lower heart rate, higher sucking rate, a more relaxed appearance, and less crying and body movements.
  Interventions: Other: Mother voice

INTERVENTIONS:
Other: Mother voice — Five minutes before the procedure, the mother's voice recording will be played to the baby and the speaker will be placed 30 cm away from the baby. The baby's comfort level will be evaluated by the researcher using the "Neonatal Comfort Behavior Scale" 2 minutes before the procedure begins. Physiological values of the baby will be noted by the researcher 1 minute before the procedure.As soon as the heel blood procedure is completed, the baby's physiological values and comfort level will be noted by the "Newborn Comfort Behavior Scale" by the researcher. After the procedure, the recording will continue to be played until the baby's mother's voice returns to the basal values. Physiological values and comfort levels of the baby will be noted by the researcher 1 minute and 2 minute after the procedure. 2 minutes after the procedure, the baby's comfort level will be evaluated by the researcher using the "Neonatal Comfort Behavior Scale".
  Arms: Mother Voice
Other: White noise — Before Operation The decibel meter will be set to an average of 50-60 dB and the speakers will be played at a distance of 30 cm.
  Intervention in this group will be made at the elevation. White noise will be played five minutes before the procedure.The baby's comfort level and physiological values will be evaluated by the researcher using the "Neonatal Comfort Behavior Scale" 2 minutes before the procedure begins.
  Order of Operation As soon as the heel blood procedure is completed, the baby's physiological values and comfort level will be noted by the "Newborn Comfort Behavior Scale" by the researcher.
  Post-Processing After the procedure, white noise will continue to be listened to until the baby's physiological values return to basal values. Physiological values and baby's comfort level of the baby will be noted by the researcher 1 minute and 2 minute after the heel blood collection is completed.
  Arms: White Noise

SUMMARY:
The heel blood procedure for newborn screening is done for almost all babies within the first 48 hours of birth. It is stated that non-pharmacological methods in reducing pain during the heel blood collection process are simple, effective, free, and very cost-effective. Studies have shown that auditory interventions (such as mother's voice, white noise) used in invasive procedures distract the infant and create a cognitive strategy for pain control. According to this information, one aim of the study is to determine the effect of the mother's voice and white noise, which are non-pharmacological methods, on the comfort level of the baby in the heel blood procedure. It is thought that especially acute painful procedures applied to infants will reduce the level of stress and anxiety in parents. Another aim of this study is to determine the effect of a mother's voice and white noise, which are non-pharmacological methods, on the state anxiety levels of mothers in the heel blood collection process.

DETAILED DESCRIPTION:
The heel blood procedure for newborn screening is done for almost all babies within the first 48 hours of birth. The heel blood procedure, which is widely used for the diagnosis and follow-up of various diseases, causes acute pain in infants. It is stated that non-pharmacological methods in reducing pain during the heel blood collection process are simple, effective, free, and very cost-effective. For example, non-pharmacological methods such as breastfeeding, skin-to-skin contact, oral sucrose, mother's voice, and white noise are stated to be effective in reducing acute pain. Clinical practice guidelines recommend the use of non-pharmacological methods in acute painful procedures. Studies have shown that auditory interventions (such as mother's voice, white noise) used in invasive procedures distract the infant and create a cognitive strategy for pain control. According to this information, one aim of the study is to determine the effect of the mother's voice and white noise, which are non-pharmacological methods, on the comfort level of the baby in the heel blood procedure.

Few studies have targeted parents of newborn infants, although studies to date have shown that parents want to be more involved in their infants' pain management. Parents reported that they wanted to learn more about pain management strategies, they wanted to play a role in the relaxation of their babies, and they hoped for more opportunities to participate in the care of their babies in the hospital. It is thought that especially acute painful procedures applied to infants will reduce the level of stress and anxiety in parents. In addition, one study reported that when parents are given information to help reduce their baby's pain, they accept painful procedures such as heel prick more easily and feel calmer. In the light of this information, another aim of this study is to determine the effect of a mother's voice and white noise, which are non-pharmacological methods, on the state anxiety levels of mothers in the heel blood collection process.

ELIGIBILITY:
Inclusion Criteria:

1. Newborns whose postnatal age is between 1-5 days,
2. 38-42. newborns born between gestational weeks,
3. Healthy newborns,
4. Babies of mothers without diabetes,
5. Newborns who were not given any opioid and non-opioid drugs before the application,
6. Newborns who have been fed at least 30 minutes ago,
7. Newborns without any painful interventions other than vitamin K and Hepatitis B injections will be included.
8. Mothers who can speak and understand Turkish,
9. The mothers and their babies who accepted to participate in the study and whose written consent form was obtained from them will be included in the study.

Exclusion Criteria:

1. Connected to a mechanical ventilator,
2. Having a neurological disorder,
3. Congenital anomaly,
4. Having hyperglycemia,
5. Having undergone a surgical procedure,
6. Substance addicted mother and her baby,
7. If the lancet cannot be inserted and removed at once, the baby will be excluded from the study.
8. Infants, despite meeting the criteria, will be excluded from the study if the heel blood collection takes more than 2 minutes in total, the procedure is disrupted by someone entering the room loudly, or the mother changes the position of the baby.
9. Mothers with a special condition that will cause difficulties in understanding and perception will be excluded from the study.

Ages: 1 Hour to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-16 (Actual)

PRIMARY OUTCOMES:
CONFORTneo Scale | 1 year
  The Neonatal Comfort Behavior Scale consists of 7 items: muscle tone, alertness, facial tension, calmness/agitation, body movements, respiratory response, and crying. Since "respiratory response" was scored in infants connected to mechanical ventilator and "crying" was scored in spontaneously breathing infants, the total score was calculated over 6 items. The lowest score that can be obtained from the Newborn Comfort Behavior Scale is 6, and the highest score is 30.On this scale, if the total score of the scale is between 6-13, the baby is comfortable. If the total score is between 14-30, the baby has pain or distress and needs interventions to relieve him.

SECONDARY OUTCOMES:
Heart rate peak | 1 year
  Peak heart rate will be measured with the "Nellcor Oximax N-560 Quick Guide" brand device. Nellcor saturation probe will be attached to the left foot of the newborn and the measurement will be made by the investigator.
Oxygen saturation | 1 year
  Oxygen saturation will be measured with the "Nellcor Oximax N-560 Quick Guide" brand device. Nellcor saturation probe will be attached to the left foot of the newborn and the measurement will be made by the investigator.
Crying time | 1 year
  The crying time of the newborn will be recorded by the researcher. Time to return to baseline values
State Anxiety Scale score | 1 year
  In this study, the "State Anxiety" section of the State-Trait Anxiety Inventory developed by Spielberg et al. in 1970 will be used to determine the state anxiety levels of mothers.
  In the evaluation, 0-19 points are interpreted as "no anxiety", 20-39 points as "mild anxiety", 40-59 points as "moderate anxiety", 60-79 points as "severe anxiety" and 80 points as "panic value".

CONTACTS AND LOCATIONS:
Overall Officials: Uğur Gül, Principal Investigator — Akdeniz Universitesi, Akdeniz University Faculty of Nursing
Locations (1):
- Akdeniz University, Kepez, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The identity of the patient will not be shared to ensure confidentiality.

REFERENCES:
- [Background] Axelin A, Anderzen-Carlsson A, Eriksson M, Polkki T, Korhonen A, Franck LS. Neonatal Intensive Care Nurses' Perceptions of Parental Participation in Infant Pain Management: A Comparative Focus Group Study. J Perinat Neonatal Nurs. 2015 Oct-Dec;29(4):363-74. doi: 10.1097/JPN.0000000000000136. PMID 26505851
- [Background] Benoit B, Campbell-Yeo M, Johnston C, Latimer M, Caddell K, Orr T. Staff Nurse Utilization of Kangaroo Care as an Intervention for Procedural Pain in Preterm Infants. Adv Neonatal Care. 2016 Jun;16(3):229-38. doi: 10.1097/ANC.0000000000000262. PMID 27148835
- [Background] Benoit B, Martin-Misener R, Latimer M, Campbell-Yeo M. Breast-Feeding Analgesia in Infants: An Update on the Current State of Evidence. J Perinat Neonatal Nurs. 2017 Apr/Jun;31(2):145-159. doi: 10.1097/JPN.0000000000000253. PMID 28437305
- [Background] Campbell-Yeo M, Fernandes A, Johnston C. Procedural pain management for neonates using nonpharmacological strategies: part 2: mother-driven interventions. Adv Neonatal Care. 2011 Oct;11(5):312-8; quiz pg 319-20. doi: 10.1097/ANC.0b013e318229aa76. PMID 22123399
- [Background] Cong X, Delaney C, Vazquez V. Neonatal nurses' perceptions of pain assessment and management in NICUs: a national survey. Adv Neonatal Care. 2013 Oct;13(5):353-60. doi: 10.1097/ANC.0b013e31829d62e8. PMID 24042143
- [Background] Cong X, McGrath JM, Delaney C, Chen H, Liang S, Vazquez V, Keating L, Chang K, Dejong A. Neonatal nurses' perceptions of pain management: survey of the United States and China. Pain Manag Nurs. 2014 Dec;15(4):834-44. doi: 10.1016/j.pmn.2013.10.002. Epub 2014 Feb 6. PMID 24508269
- [Background] Franck LS, Oulton K, Bruce E. Parental involvement in neonatal pain management: an empirical and conceptual update. J Nurs Scholarsh. 2012 Mar;44(1):45-54. doi: 10.1111/j.1547-5069.2011.01434.x. Epub 2012 Feb 16. PMID 22339845
- [Background] Harrison D, Larocque C, Bueno M, Stokes Y, Turner L, Hutton B, Stevens B. Sweet Solutions to Reduce Procedural Pain in Neonates: A Meta-analysis. Pediatrics. 2017 Jan;139(1):e20160955. doi: 10.1542/peds.2016-0955. Epub 2016 Dec 16. PMID 27986905
- [Background] Karakoc A, Turker F. Effects of white noise and holding on pain perception in newborns. Pain Manag Nurs. 2014 Dec;15(4):864-70. doi: 10.1016/j.pmn.2014.01.002. Epub 2014 Feb 20. PMID 24559599
- [Result] Kahraman A, Gumus M, Akar M, Sipahi M, Bal Yilmaz H, Basbakkal Z. The effects of auditory interventions on pain and comfort in premature newborns in the neonatal intensive care unit; a randomised controlled trial. Intensive Crit Care Nurs. 2020 Dec;61:102904. doi: 10.1016/j.iccn.2020.102904. Epub 2020 Jul 9. PMID 32653359